CLINICAL TRIAL: NCT07154134
Title: Comparative Study Between Endocan and Copeptin Serum Levels in Preterm Neonates With Respiratory Distress Syndrome
Brief Title: Endocan and Copeptin Serum Levels in Preterm Neonates With Respiratory Distress Syndrome
Status: Recruiting | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Asmaa Mahmoud Abdel Hamid Elmesiry, Lecturer of Pediatrics, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Other Study IDs: 36264PR1296/7/25
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Endocan; Copeptin; Serum; Preterm Neonates; Respiratory Distress Syndrome
MeSH Terms: conditions — Diabetes Insipidus; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: Neonates with gestational ages between 28 and 34 gestational weeks.
  Interventions: Diagnostic Test: Serum endocan; Diagnostic Test: Serum copeptin
- Group II: Neonates with gestational ages between 34 and 36 gestational weeks.
  Interventions: Diagnostic Test: Serum endocan; Diagnostic Test: Serum copeptin

INTERVENTIONS:
Diagnostic Test: Serum endocan — Serum endocan will be measured by an enzyme-linked immunosorbent assay (ELISA) on the first day of life.
Diagnostic Test: Serum copeptin — Serum copeptin will be measured by an enzyme-linked immunosorbent assay (ELISA) on the first day of life.

SUMMARY:
This work aims to investigate and compare the levels of serum endocan and serum copeptin on the first day of life and correlate their levels to the severity of respiratory distress in preterm neonates suffering from respiratory distress syndrome.

DETAILED DESCRIPTION:
Preterm birth continues to be one of the significant challenges in perinatal medicine because of its high incidence of morbidities and mortalities. Its burden on the infant, the family, healthcare systems, and society is enormous.

Endocan is implicated in the recruitment of circulating lymphocytes to inflammatory sites and leukocyte adhesion and activation. Endocan also inhibits leukocyte-endothelial cell adhesion and reduces the excessive leukocyte recruitment into the lungs.

Copeptin, also known as the arginine vasopressin (AVP) associated glycopeptides. AVP is a vasoactive neurohypophysial hormone. It is one of the primary hormones of the hypothalamic-pituitary-adrenal axis, and its primary function is to regulate water and maintain electrolyte homeostasis. The primary stimulus for AVP release is hyperosmolarity.

ELIGIBILITY:
Inclusion Criteria:

* Prematurity.
* Gestational age between 28 and 36 weeks.
* Suffering from respiratory distress syndrome.

Exclusion Criteria:

* Intrauterine growth restriction (IUGR).
* Hypoxic ischemic encephalopathy.
* Multiple congenital anomalies.
* Chromosomal abnormalities.
* Preterm less than 28 weeks.
* Neonates with a maternal history of chorioamnionitis (early sepsis).
* Infant of diabetic mother.
* Prelabor rupture of membranes (PROM)> 2 hours.

Ages: 28 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This prospective study will be conducted at the Neonatal Intensive Care Unit (NICU), Pediatric Department, Tanta University Hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Serum endocan level for prediction of severity of respiratory distress syndrome | First day of life
  Serum endocan level for prediction of severity of respiratory distress syndrome (RDS) will be recorded.

SECONDARY OUTCOMES:
Serum copeptin level for prediction of severity of respiratory distress syndrome | 5th day of life
  Serum copeptin level for the prediction of the severity of respiratory distress syndrome (RDS) will be recorded.
Serum endocan level for prediction of mortality | First day of life
  Serum endocan level for prediction of mortality will be recorded.
Serum copeptin level for prediction of mortality | 5th day of life
  Serum copeptin level for prediction of mortality will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.